CLINICAL TRIAL: NCT00262769
Title: Gemcitabine, Alone or in Combination With Cisplatin, in Patients With Advanced or Metastatic Cholangiocarcinomas and Other Biliary Tract Tumors: A Multicentre, Randomized Phase III Study
Brief Title: Gemcitabine With or Without Cisplatin in Treating Patients With Unresectable Locally Advanced or Metastatic Cholangiocarcinoma or Other Biliary Tract Tumors
Acronym: ABC-02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000455013; CRUK-ABC-02; EU-205103; ISRCTN82956140; EUDRACT-2004-004882-14; CTA-21266/0005/001
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer
Keywords: cholangiocarcinoma of the extrahepatic bile duct; recurrent extrahepatic bile duct cancer; unresectable extrahepatic bile duct cancer; cholangiocarcinoma of the gallbladder; recurrent gallbladder cancer; unresectable gallbladder cancer; metastatic extrahepatic bile duct cancer; metastatic gallbladder cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A - Gemcitabine (Experimental): Gemcitabine alone
  Interventions: Drug: gemcitabine hydrochloride
- B - Gemcitabine and Cisplatin (Experimental): Gemcitabine and Cisplatin
  Interventions: Drug: cisplatin; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: cisplatin — 25 mg/m2 in 1000 mls 0.9% saline given over 1 hour followed by 500 mls 0.9% saline over 90 mins
  Other Names: CDDP; cis-diamminedichloroplatinum(II); cisplatinum
  Arms: B - Gemcitabine and Cisplatin
Drug: gemcitabine hydrochloride — 1000mg/m2 in 250-500mls 0.9% saline over 30 mins by intravenous infusions on day 1, 8 and 15 (Arm A only) of each 28 (Arm A) or 21 (Arm B) day cycle.
  Other Names: Gemzar

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known whether gemcitabine is more effective with or without cisplatin in treating cholangiocarcinoma or biliary tract tumors.

PURPOSE: This randomized phase III trial is studying gemcitabine and cisplatin to see how well they work compared to gemcitabine alone in treating patients with unresectable locally advanced or metastatic cholangiocarcinoma or other biliary tract tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of patients with unresectable locally advanced or metastatic cholangiocarcinoma or other biliary tract tumors treated with gemcitabine hydrochloride with vs without cisplatin.

Secondary

* Compare the progression-free survival of patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.
* Compare quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, primary site of disease (gallbladder vs bile ducts vs ampulla), prior therapy (photodynamic therapy [PDT] vs non-PDT therapy vs none), ECOG performance status (0 vs 1 vs 2), and disease status (locally advanced vs metastatic). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive gemcitabine hydrochloride IV over 30 minutes and cisplatin IV over 1½ hours on days 1 and 8. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, 12 weeks, and after finishing treatment.

After completion of study treatment, patients are followed periodically for at least 3 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 400 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed biliary tract, gallbladder, or ampullary carcinoma

  * Intra- or extra-hepatic disease allowed
* Unresectable locally advanced, recurrent, or metastatic disease
* No brain metastases

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL (transfusion allowed)
* WBC ≥ 3,000/mm^3

Hepatic

* AST and ALT ≤ 3 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Bilirubin ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 3 times ULN (5 times ULN if liver metastases are present)
* Adequate biliary drainage
* No unresolved biliary tract obstruction

Renal

* Creatinine < 1.5 times ULN
* Urea < 1.5 times ULN
* Glomerular filtration rate (GFR) ≥ 45 mL/min

  * If GFR < 60 mL/min, isotope EDTA confirmation of adequate renal function is required

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No active, uncontrolled infection
* No other severe or uncontrolled systemic disease
* No other malignancy within the past 5 years except nonmetastatic basal cell or squamous cell skin cancer or carcinoma in situ of the cervix treated by cone-biopsy or resection
* No psychiatric disorder that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

Chemotherapy

* At least 6 months since prior adjuvant chemotherapy
* No prior gemcitabine hydrochloride
* No prior cisplatin
* No prior systemic chemotherapy for locally advanced or metastatic disease except low-dose radiosensitizing chemotherapy in conjunction with radiotherapy

Radiotherapy

* Prior radiotherapy for localized disease allowed provided there is clear evidence of disease progression afterwards

Surgery

* Prior curative surgery allowed provided there is evidence of nonresectable disease relapse requiring systemic chemotherapy

Other

* Recovered from all prior therapies
* Prior photodynamic therapy (PDT) allowed provided it was given for localized disease only (with no evidence of metastatic disease) and resulted in subsequent disease progression after completion of therapy OR to relieve biliary obstruction in the presence of metastatic disease

  * PDT must have been completed ≥ 4 weeks ago
* At least 4 weeks since prior investigational agents
* No other concurrent, curative anticancer therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2005-05; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From date of randomisation till date of death or last date of follow-up (up to 5 years)
  From date of randomisation till date of death or last date of follow-up (up to 5 years)

SECONDARY OUTCOMES:
Progression-free survival | From date of randomisation till date of death or last date of follow-up (up to 5 years)
  From date of randomisation till date of death or last date of follow-up (up to 5 years)
Quality of life | Before and 12 weeks after completion of treatment
  Quality of life as measured by EORTC Quality of Life Questionnaire Core 30 Items periodically
Toxicity | During treatment and follow-up
  Toxicity as measured by NCI CTC periodically. The proportion of patients who experience a toxicity of grade 3 or 4 will be compared between the two arms of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: John A. Bridgewater, Study Chair — University College London (UCL) Cancer Institute
Locations (25):
- United Kingdom (25):
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Addenbrooke's Hospital, Cambridge, England
  - Cumberland Infirmary, Carlisle, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Derbyshire Royal Infirmary, Derby, England
  - Princess Alexandra Hospital, Essex, England
  - Gloucestershire Royal Hospital, Gloucester, England
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Helen Rollason Cancer Care Centre at North Middlesex Hospital, London, England
  - Royal Marsden - London, London, England
  - Hammersmith Hospital, London, England
  - UCL Cancer Institute, London, England
  - University College of London Hospitals, London, England
  - Maidstone Hospital, Maidstone, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital, Nottingham, England
  - Portsmouth Oncology Centre at Saint Mary's Hospital, Portsmouth Hants, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Belfast City Hospital Trust Incorporating Belvoir Park Hospital, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales

REFERENCES:
- [Result] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404